CLINICAL TRIAL: NCT04273321
Title: Efficacy and Safety of Corticosteroids in COVID-19: A Prospective Randomized Controlled Trails
Brief Title: Efficacy and Safety of Corticosteroids in COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Shi Huanzhong, Professor, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Methylprednisolone in COVID-19
Record Dates: First submitted 2020-02-15; First posted 2020-02-18 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; Novel Coronavirus Pneumonia
MeSH Terms: conditions — COVID-19 | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MP group (Experimental)
  Interventions: Drug: Methylprednisolone
- Con group (No Intervention)

INTERVENTIONS:
Drug: Methylprednisolone — Methylprednisolone 1mg/kg/day ivgtt for 7 days.
  Arms: MP group

SUMMARY:
There is still controversy about the effective of glucocorticoids for the treatment of novel coronavirus pneumonia. This is a prospective randomized controlled trails. The aim is to explore the effectiveness and safety of glucocorticoids in the treatment of novel coronavirus pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years old
* accord with the clinical diagnosis and/ or etiological diagnosis diagnostic criteria of Novel coronavirus pneumonia (COVID-19).
* admitted in the general wards
* be able to sign informed consent

Exclusion Criteria:

* severe immunosuppression (HIV infection, long-term use of immunosuppressive agents
* pregnant or lactation period women
* glucocorticoids are needed for other diseases
* unwilling or unable to participate or complete the study
* participate in other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
the incidence of treatment failure in 14 days | 14 days
  The clinical symptoms and signs continue to deteriorate, or new pulmonary or extrapulmonary lesions appear, or the chest imaging indicates the progress, and the patient is transferred to ICU or intubation and invasive ventilation or died.

SECONDARY OUTCOMES:
clinical cure incidence in 14 days | 14 days
  The clinical symptoms and signs improved or alleviated (the temperature be normal , respiratory symptoms improved significantly, imaging showed obvious absorption) and no additional or alternative treatment was needed.
the duration of virus change to negative | 30 days
  the duration from admission to virus negative
mortality at day 30 | 30 days
  the patient die in 30 days
ICU admission rate in 30 days | 30 days
  the patients transform to ICU because of clinical deteriorate in 30 days

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Hubei province hospital of integrated Chinese & Western Medicine, Wuhan, Hubei
  - Yichang first people's Hospital, Yichang, Hubei
  - Beijing YouAn Hospital, Beijing
  - Renmin Hospital of Wuhan University, Wuhan
  - Tianyou Hospital Affiliated to Wuhan University of science and technology, Wuhan
  - Union Hospital Affiliated to Tongji Medical College of Huazhong University of science and technology, Wuhan
  - the first peopel hospital of Xiangyang, Xiangyang

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

REFERENCES:
- [Derived] Tang X, Feng YM, Ni JX, Zhang JY, Liu LM, Hu K, Wu XZ, Zhang JX, Chen JW, Zhang JC, Su J, Li YL, Zhao Y, Xie J, Ding Z, He XL, Wang W, Jin RH, Shi HZ, Sun B. Early Use of Corticosteroid May Prolong SARS-CoV-2 Shedding in Non-Intensive Care Unit Patients with COVID-19 Pneumonia: A Multicenter, Single-Blind, Randomized Control Trial. Respiration. 2021;100(2):116-126. doi: 10.1159/000512063. Epub 2021 Jan 22. PMID 33486496